CLINICAL TRIAL: NCT02906163
Title: First Line Bio-immunotherapy With Thymosin Alpha 1 in Patients With Sensitizing EGFR Mutation Positive Non Small Cell Lung Cancer Who Are Taking Standard of Care Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI-Ta1-NSCLC-P1/2-001
Record Dates: First submitted 2016-08-29; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: EGFR Mutation Positive Non Small Cell Lung Cancer
Keywords: EGFR mutation positive; Thymosin Alpha 1; Tyrosine Kinase inhibitor; Thymalfasin; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thymalfasin; Trace amine-associated receptor 1; Tyrosine Kinase Inhibitors; Afatinib; Gefitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Thymalfasin biw plus SoC (tyrosine kinase inhibitor) (Experimental): Twice weekly thymalfasin
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1); Drug: SoC (tyrosine kinase inhibitor)
- Thymalfasin plus SoC (tyrosine kinase inhibitor) (Experimental): 5 times a week thymalfasin
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1); Drug: SoC (tyrosine kinase inhibitor)
- SoC (tyrosine kinase inhibitor) (Active Comparator): 12 months
  Interventions: Drug: SoC (tyrosine kinase inhibitor)

INTERVENTIONS:
Drug: Thymalfasin (Thymosin alpha 1, Ta1) — In Phase I patients will be randomized to one of two different dosing regimens of Thymosin alpha 1 for a treatment duration of 4 months. At the completion of Phase I, data will be reviewed and a single dosing regimen will be carried forward into Phase II.
  Other Names: ZADAXIN
  Arms: Thymalfasin biw plus SoC (tyrosine kinase inhibitor); Thymalfasin plus SoC (tyrosine kinase inhibitor)
Drug: SoC (tyrosine kinase inhibitor) — In Phase II patients will be randomized to SoC or Thymosin alpha 1 plus SoC for treatment duration of 12 months. All patients will be followed for approximately 18 months.
  Other Names: afatinib, gefitinib, erlotinib

SUMMARY:
Phase I: evaluate the safety and tolerability two different dosing regimens of Thymosin alpha 1 in patients with advanced EGFR mutation positive NSCLC on Standard of Care (SoC) therapy.

Phase II: evaluate the efficacy in terms of PFS of Thymosin alpha 1 in patients with advanced EGFR mutant NSCLC taking SoC as compared to SoC alone.

DETAILED DESCRIPTION:
Phase I/Phase II, multi-center, open label, randomized, parallel group study to determine the safety/tolerability/efficacy of Thymosin alpha 1 in patients with sensitizing EGFR mutation positive NSCLC taking SoC versus SoC alone. The study will be conducted in subjects with sensitizing EGFR mutation positive Non Small Cell Lung Cancer. Subjects with sensitizing EGFR mutation positive NSCLC will be screened for eligibility by the clinical center involved. The study will be conducted in two parts. In Phase I patients will be randomized to one of two different dosing regimens of Thymosin alpha 1 for a treatment duration of 4 months. At the completion of Phase I, data will be reviewed and a single dosing regimen will be carried forward into Phase II. In Phase II patients will be randomized to SoC or Thymosin alpha 1 plus SoC for treatment duration of 12 months. All patients will be followed for approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histological or cytological confirmation of NSCLC (may be from initial diagnosis of NSCLC or subsequent biopsy). Only patients with available tissue samples may be included in the study (see major details in section 8 for the minimum sample characteristics)
* Activating mutations of EGFRdiagnosis of Stage IIIB (with cytologically proven pleural effusion or pericardial effusion) or metastaticNSCLC, not amenable to curative surgery or radiotherapy
* Measurable disease by Response Evaluation Criteria In Solid Tumours (RECIST) in a lesion not previously irradiated or non-measurable disease (non measurable disease only for Phase I)
* Eastern Cooperative Oncology Group - performance status (ECOG-PS) 0-2
* Absolute neutrophil count (ANC) > 1.5 x 109/liter (L) and platelets > 100 x 109/L
* Bilirubin level either normal or <1.5 x ULN
* AST (SGOT) and ALT (SGPT) <2.5 x ULN (≤ 5 x ULN if liver metastases are present)
* Serum creatinine <1.5 x ULN
* Effective contraception for both, male and female patients, if the risk of conception exists
* Provision of written informed consent to the analysis of biological markers (registration)

Exclusion Criteria:

* Prior therapy with Thymosin alpha-1
* Prior chemotherapy for relapsed and/or metastatic NSCLC. Neoadjuvant/adjuvant chemotherapy is permitted if at least 12 months has elapsed between the end of chemotherapy and randomisation.
* Prior treatment with Epidermal Growth Factor Receptor targeting small molecules or antibodies
* Radiotherapy within 14 days prior to drug administration, except as follows:
* Palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
* Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically stable disease (SD) (no steroid therapy or steroid dose being tapered) for at least 28 days
* Patients with toxicities that have not coming back (at least) to grade 1
* Pregnancy or suspected pregnancy
* Known severe hypersensitivity to TKI
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any evidence of clinically active interstitial lung disease (ILD) (patients with chronic, stable, radiographic changes who are asymptomatic or patients with uncomplicated progressive lymphangitic carcinomatosis need not be excluded)
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* As judged by the investigator, any inflammatory changes of the surface of the eye
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related adverse events | Up to 4 months
PFS | Up to12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Paolo Marchetti, MD, Principal Investigator — S. Andrea Hospital
Locations (5):
- Italy (5):
  - Azienda Sanitaria Locale Frosinone, Frosinone
  - Istituto Nazionale dei Tumori, Milan
  - Roma_Campus Bio-Medico, Rome
  - Sant'Andrea Hospital, Rome
  - Presidio Sanitario San Camillo, Torino

IPD SHARING:
Plan to Share IPD: Undecided